CLINICAL TRIAL: NCT05591716
Title: Evaluation of the Efficacy and Safety of Unimodal Bilateral Flexible Ureteroscopy A Prospective Multicenter Study
Brief Title: Evaluation of the Efficacy and Safety of Unimodal Bilateral Flexible Ureteroscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, nariman.gadjiev, Ph.D., Deputy Director for medical care (urology), Urologist of Saint Petersburg State University Clinic of advanced medical technologies n.a. N.I.Pirogov., Saint Petersburg State University, Russia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni_or_bilateral
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Kidney Stone
Keywords: urolithias; flexible urethroscopy; bilateral flexible urethroscopy; lazer
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral flexible ureteroscopy (Active Comparator): Transurethral removal of kidney stones
  Interventions: Procedure: Unilateral same-session flexible ureterorenoscopy
- Bilateral flexible ureteroscopy (Active Comparator): Transurethral removal of kidney stones
  Interventions: Procedure: Bilateral same-session flexible ureterorenoscopy

INTERVENTIONS:
Procedure: Bilateral same-session flexible ureterorenoscopy — The patient was in the lithotomic position. A semi-rigid ureteroscope was passed into the bladder, then a roadrunner was placed. A flexible urethroscope is guided along the roadrunner to the kidney. In the kidney, the concrement is fragmented with laser energy. The fragments were extracted using a basket. Then a revision of the kidney is performed using a flexible urethroscope. A ureteral stent was placed in the pelvis.The ureteroscope was extracted together with the case with the ureteral revision: there was no damage to the ureter.Next, this procedure is performed from the other side. Urine was excreted from the bladder using a Nelaton catheter.
  Arms: Bilateral flexible ureteroscopy
Procedure: Unilateral same-session flexible ureterorenoscopy — The patient was in the lithotomic position. A semi-rigid ureteroscope was passed into the bladder, then a roadrunner was placed. A flexible urethroscope is guided along the roadrunner to the kidney. In the kidney, the concrement is fragmented with laser energy. The fragments were extracted using a basket. Then a revision of the kidney is performed using a flexible urethroscope. A ureteral stent was placed in the pelvis. The ureteroscope was extracted together with the body with revision of the ureter: there was no damage to the ureter. Urine was excreted from the bladder using a Nelaton catheter.
  Arms: Unilateral flexible ureteroscopy

SUMMARY:
This is a prospective controlled study to compare the efficacy and safety of two methods of flexible urethroscopy in patients with urolithiasis, as well as the effect of surgery on quality of life.

DETAILED DESCRIPTION:
Retrograde flexible URS is the most modern and safe method of treating patients with bowel stones up to 20 mm. Bilateral kidney stones can be treated with bilateral retrograde flexible URS. This type of surgery allows a patient to get rid of both kidney stones in a single intervention. Technically, the operation can be performed alternately on each side or simultaneously by two surgeons if two flexible instruments and video endoscopic racks are available simultaneously. Flexible ureteroscope diameter of 7.5-9 Сh enables to place two instruments even in the male urethra simultaneously without significant traumatization. One of the disadvantages of this method is the need for bilateral prestenting, with the frequency and the frequency and severity of stent-associated symptoms may increase. Few scientific works demonstrate contradictory data concerning the safety of bilateral flexible URS; therefore, further research is advisable.

All patients meeting the selection criteria will undergo preoperative examination: history, physical, laboratory and CT scan of the kidneys.

MATERIALS AND METHODS To calculate the sample, the investigators used the method for "no lesser efficiency" studies. To confirm the hypothesis of no greater number of complications in the form of upper urinary tract mucosal damage, exit (extravasation) of irrigation solution outside the upper urinary tract, bleeding and perforation of the ureteral wall, which according to the literature are 11.9% for bilateral and 8.5% for unilateral RIRH respectively, a minimum of 82 patients would be required in order to study of 80% and a probability of first-order error of 5% to exclude a 20% difference in the number of complications, which is clinically significant. To compensate for data loss, the sample size is increased by 5% to 86 patients. Categorical variables will be reported as absolute numbers and percentages. Unadapted univariate analyses, to compare the two treatment groups, will be based on Fisher's exact test. Relative risks and 95% confidence intervals will be calculated using the two-by-two table method using a logarithmic approximation. Continuous variables will be displayed as mean ± standard deviation or median and interquartile range.Pre- and postoperative data collected will be anonymized using unique codes that patients will receive immediately after randomization.

All surgical procedures will be performed by 3 qualified surgeons. Postoperative follow-up will be performed 1 day,1 month after surgery by two investigators, a non-blinded study.

ELIGIBILITY:
Inclusion Criteria:

* Single and bilateral kidney stones with a total 20 mm or less on each side
* Over 18 years of age
* Signed informed consent

Exclusion Criteria:

* Patients with large stones (total size greater than 20 mm) and coral stones
* Urethral and ureteral strictures
* Urinary tract abnormalities
* Unwillingness to sign informed consent
* Presence of active urinary tract infection
* Pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-02-17 (Estimated); Study Completion 2023-05-17 (Estimated)

PRIMARY OUTCOMES:
Objective cure rate | 1 day after surgery surgery
  The frequency of early postoperative complications according to Clavien-Dindo scale starting from the second stage more.

SECONDARY OUTCOMES:
Assessment of kidney performance | 1 day after surgery surgery
  Assessment of plasma creatinine level
Assessment of the inflammatory process | 1 day after surgery surgery
  body temperature
Postoperative examination | 1 day after surgery surgery
  Leukocyte count
Evaluation residual stones | 1 month after surgery surgery
  Hydronephrosis and residual stones according to according to ultrasound of kidneys
Evaluation stone free rate | 3 month after surgery surgery
  CT scan kidneys

CONTACTS AND LOCATIONS:
Overall Officials: Nariman Gadjiev, PhD, Study Chair — Saint Petersburg State University Hospital
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia